CLINICAL TRIAL: NCT06366802
Title: Cohort Construction and Prognostic Model Construction for Multiple Myeloma
Status: Active, not recruiting | Type: Observational
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: Prognosis model-MM09
Record Dates: First submitted 2024-02-01; First posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multiple myeloma (MM) is a disease caused by malignant plasma cell proliferation disorder. Survival outcomes continue to vary widely even within uniformly treated clinical trial populations. How to construct a clinical prognosis model of MM through real-world data to guide the selection of treatment options, standardize patient management, and improve survival expectations, is a major problem that needs to be solved urgently. It is necessary to build an MM-specific cohort in China to comprehensively understand the characteristics of MM patients, explore treatment options, and improve prognostic factors for survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients were diagnosed as multiple myeloma from January 1, 2008 (the diagnostic criteria are based on "Chinese Guidelines for the Diagnosis and Treatment of Multiple Myeloma (Revised in 2020)").

Exclusion Criteria:

Long-term follow-up information for patients is not available for any reason, such as not being available or having a serious concomitant disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Newly diagnosed MM patients admitted to the First Affiliated Hospital of Soochow University
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2027-05-02 (Estimated); Study Completion 2027-05-02 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Overall survival is defined as the time from being treated to death from any cause.

SECONDARY OUTCOMES:
Progression free survival(PFS) | 5years
  Progression-free survival (PFS) is defined as the time from being treated to disease progression or death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China